CLINICAL TRIAL: NCT06054854
Title: Biobank for the Identification of Diagnostic, Prognostic or Therapeutic (Response and Resistance) Biomarkers in Lung Cancer (Early and Advanced Stages of Lung Cancer Cohort of the BIRD (Biomarkers in Respiratory Disease) Biobank)
Brief Title: Biobank for the Identification of Biomarkers in Lung Cancer (BIRD, Biomarkers in Respiratory Disease)
Acronym: BIRD-NK
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0492
Record Dates: First submitted 2023-09-07; First posted 2023-09-26 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Lung Nodule; Lung Cancer
Keywords: Lung Nodule; Lung Cancer; Early Stage Lung Cancer; Advanced Lung Cancer; Liquid Biopsy; Biomarkers
MeSH Terms: conditions — Lung Neoplasms | interventions — Medical Waste

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extra blood sampling. Urine, Saliva, Stool, Superficial nasal swamp sampling. Bronchoalveolar lavage fluid, Mediastinal node or mass, Peripheral nodule aspiration supernatant, Pleural fluid, Cerebrospinal fluid collection (leftover samples or medical waste).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with lung nodule or lung cancer: Patients suspected of or suffering from early stage (supracentimetric nodule) or advanced thoracic cancer
  Interventions: Biological: Extra blood sampling, Non-invasive or leftover samples or medical waste

INTERVENTIONS:
Biological: Extra blood sampling, Non-invasive or leftover samples or medical waste — Extra blood sampling, Urine, Saliva, Stool, Superficial nasal swamp sampling. Bronchoalveolar lavage fluid, Mediastinal node or mass, Peripheral nodule aspiration supernatant, Pleural fluid, Cerebrospinal fluid collection (leftover samples or medical waste).
  Blood will be collected in larger quantity during a blood test planned as part of the patient's care.
  Non-invasive or leftover samples or medical waste will be collected on top of the usual diagnosis and during follow-up, depending on the case.

SUMMARY:
The BIRD biobank aims at collecting clinical and biological data from patients suffering from a chronic respiratory disease. The lung cancer subpopulation will be divided into two cohorts to identify biomarkers of cancer. One cohort will include patients with supra-centimetric lung nodule(s) whether surveillance, bronchoscopic or radio-guided biopsy or surgery is indicated, patients suspected of lung cancers requiring diagnostic and/or therapeutic bronchial endoscopy and patients with a known early stage lung cancer (early-stage cohort). The second cohort will include known advanced stage lung cancers (III-IV).

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death. In France, lung cancer is a common cancer (fourth cause of cancer) with 49,000 new cases diagnosed each year and nearly 29,000 deaths per year.

New therapies (targeted therapies and immune checkpoint inhibitors) are now available and improve patient care. However, their prescription is based on the molecular analysis of the biopsies which are often of very small size, sometimes performed on lesions that are difficult to access, requiring invasive sampling that are difficult to repeat over time.

Identifying biomarkers via different fluids that are easier to access (blood, bronchiolo-alveolar lavage, etc.) therefore is strongly needed to improve screening and diagnosis and to optimize treatment.

The objectives of this biobank are:

To identify diagnostic, theragnostic, prognostic or therapeutic biomarkers in early and advanced stage lung cancer.

To evaluate the prevalence of lung cancer and identify predictive biomarkers for malignancy in patients with lung nodule(s).

To test the feasibility and diagnostic yield of the detection of known biomarkers in non or less invasive biological specimens (blood, urine, other) and analyse the concordance with tissue biopsy.

To identify mechanisms of oncogenesis and identify new molecular targets for anticancer treatment using genomics, transcriptomics or proteomics.

After informed consent, clinical data and biological samples will be collected up to 15 years, at the inclusion of the patients in the cohort, and at each monitoring programmed in their usual care. Up to 10 different biological fluids (blood (up to 55 ml), bronchoalveolar lavage, mediastinal node or mass, or peripheral nodule aspiration supernatant, urine, pleural fluid, cerebrospinal fluid, saliva, nasal swamp, stool) will be obtained depending on the case.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 1 to 3 lung nodules including one > 1 cm seen on chest CT
* OR: patients with suspected lung cancer requiring diagnostic and/or therapeutic bronchial endoscopy
* OR: Patient with histologically confirmed lung cancer, whether early stages prior to surgery, locally advanced or metastatic, included before the start of any anti-cancer treatment.
* Patient affiliated or beneficiary of a social security scheme
* Patients who are able to receive and understand information about the study and their participation and who have freely given their signed inform consent before any collection of samples or data necessary for the research (no restriction of rights by the judicial authorities and knowledge of the French language).

Exclusion Criteria:

* Patient deprived of liberty on administrative or judicial decision, or patient under guardianship, curators or safeguard of justice
* Female patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with lung nodule or lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2033-10-01 (Estimated); Study Completion 2033-10-01 (Estimated)

PRIMARY OUTCOMES:
Constitution of a clinico-biological collection from patients suspected of or suffering from early stage (supracentimetric nodule) or advanced thoracic cancer. | At the inclusion and up to 15 years after the inclusion
  Extra sample of blood and up to 9 different biological fluids (Urine, Saliva, Stool, Superficial nasal swamp, Bronchoalveolar lavage fluid, Mediastinal node or mass, Peripheral nodule aspiration supernatant, Pleural fluid, Cerebrospinal fluid) will be collected.

SECONDARY OUTCOMES:
Identify new biomarkers and/or sets of biomarkers in patients with lung nodules (diagnostic biomarkers) or advanced lung cancer (prognostic or therapeutic biomarkers). | At the inclusion and up to 15 years after the inclusion
  Extra sample of blood and up to 9 different biological fluids (Urine, Saliva, Stool, Superficial nasal swamp, Bronchoalveolar lavage fluid, Mediastinal node or mass, Peripheral nodule aspiration supernatant, Pleural fluid, Cerebrospinal fluid) will be collected
Explore whether known tumor markers of interest can be found in other biological samples that are easier to access (urine, blood, etc.). | At the inclusion and up to 15 years after the inclusion
  Extra sample of blood and up to 9 different biological fluids (Urine, Saliva, Stool, Superficial nasal swamp, Bronchoalveolar lavage fluid, Mediastinal node or mass, Peripheral nodule aspiration supernatant, Pleural fluid, Cerebrospinal fluid) will be collected
Estimate the concordance of the presence of known and/or newly identified biomarkers of interest in the biological sample(s) of the collection with the tissue biopsy data. | At the inclusion and up to 15 years after the inclusion
  Extra sample of blood and up to 9 different biological fluids (Urine, Saliva, Stool, Superficial nasal swamp, Bronchoalveolar lavage fluid, Mediastinal node or mass, Peripheral nodule aspiration supernatant, Pleural fluid, Cerebrospinal fluid) will be collected
Study the evolution over time of the biomarkers of interest and/or newly identified in the biological sample(s) constituting the collection. | At the inclusion and up to 15 years after the inclusion
  Extra sample of blood and up to 9 different biological fluids (Urine, Saliva, Stool, Superficial nasal swamp, Bronchoalveolar lavage fluid, Mediastinal node or mass, Peripheral nodule aspiration supernatant, Pleural fluid, Cerebrospinal fluid) will be collected
Explore through molecular and/or genomic and/or transcriptomic and/or proteomic studies the biological mechanisms underlying the development of thoracic cancer to improve screening, diagnosis, therapeutic orientation. | At the inclusion and up to 15 years after the inclusion
  Extra sample of blood and up to 9 different biological fluids (Urine, Saliva, Stool, Superficial nasal swamp, Bronchoalveolar lavage fluid, Mediastinal node or mass, Peripheral nodule aspiration supernatant, Pleural fluid, Cerebrospinal fluid) will be collected
Determine the prevalence of bronchial cancer in patients with supracentimetric lung nodules. | At the inclusion and up to 15 years after the inclusion
  Extra sample of blood and up to 9 different biological fluids (Urine, Saliva, Stool, Superficial nasal swamp, Bronchoalveolar lavage fluid, Mediastinal node or mass, Peripheral nodule aspiration supernatant, Pleural fluid, Cerebrospinal fluid) will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GUIBERT, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Larrey Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No